CLINICAL TRIAL: NCT06833203
Title: Effectiveness of Adding Amantadine to Pregabalin on Occurrence of Post-thoracotomy Pain Syndrome; Randomized Controlled Study
Brief Title: Adding Amantadine to Pregabalin on Occurrence of Post-thoracotomy Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samuel Bekhet Moawad, Assistant Lecturer of Anesthesia, Intensive Care and Pain Medicine, Faculty of Medicine, Cairo University, Cairo, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AP2310-201-002
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Amantadine; Pregabalin; Post-thoracotomy Pain Syndrome
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amantadine group (Experimental): Two hours preoperative, patient will receive two capsules, one of them is Amantadine (Amantadine Hydrochloride) 100 mg and the other is Pregabalin (Lyrica) 75 mg and continued on both of them twice daily for 5 days postoperative.
  Interventions: Drug: Amantadine+ Pregabalin
- Placebo group (Placebo Comparator): Two hours preoperative, the patient will receive two capsules, one of them is pregabalin 75 mg, and the other is a placebo capsule similar to the amantadine capsule and continued on both of them twice daily for 5 days postoperative.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Amantadine+ Pregabalin — Two hours preoperative, patient will receive two capsules, one of them is Amantadine (Amantadine Hydrochloride) 100 mg and the other is Pregabalin (Lyrica) 75 mg and continued on both of them twice daily for 5 days postoperative.
  Arms: Amantadine group
Drug: Pregabalin — Two hours preoperative, the patient will receive two capsules, one of them is pregabalin 75 mg, and the other is a placebo capsule similar to the amantadine capsule and continued on both of them twice daily for 5 days postoperative.
  Arms: Placebo group

SUMMARY:
This study aims to evaluate the additive effect of Amantadine to Pregabaline in the development of post-thoracotomy pain syndrome.

DETAILED DESCRIPTION:
Lung cancer is still the most common cause of cancer-related deaths, and lung resection surgeries could be the primary therapeutic option. Hence, the number of thoracotomy procedures is progressively increasing, as well as the development of post-thoracotomy pain syndrome (PTPS).

Pregabalin is one of the drugs that can reduce the excitability of the dorsal horn neurons. It is a γ-aminobutyric acid analogue that binds to α2-δ subunits of the voltage-gated calcium channels in the central nervous system.

Amantadine (1-aminoadamantane) is NMDA receptor antagonists. NMDA receptors were found to have role in the development of central sensitization, acute opioid tolerance, and opioid induced hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-65) years.
* Both sexes.
* American Society of Anesthesiologists (ASA) Physical status II, III.
* Body mass index (BMI): (20-40) kg/m2.
* Cancer patients undergoing posterolateral thoracotomy incision for cancer lung, mesothelioma or other lung resection procedures.

Exclusion Criteria:

* Patients with known sensitivity or contraindication to drug used in the study.
* History of psychological disorders and/or chronic pain and drug abuse patients.
* Previous administration of antidepressants, anticonvulsants, or opioids before surgery.
* Patient refusal.
* Severe respiratory or cardiac disorders.
* Advanced liver or kidney disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of occurrence of post-thoracotomy pain syndrome | 12 weeks postoperatively
  Incidence of occurrence of post-thoracotomy pain syndrome at 12 weeks through according to grading system for neuropathic pain (GSNP). GSNP is as follows: Grade 1 (unlikely), Grade 2 (possible), Grade 3 (probable), and Grade 4 (definite), the patients will be considered positive regarding incidence being in grade 3 or 4.

SECONDARY OUTCOMES:
Patient's Quality of life | 12 weeks postoperatively
  Patient's Quality of life according to Flanagan Quality of Life Scale (QOLS) which is a 16-item (domain) questionnaire with each item scored from 1 to 7 points. Participants respond to the questions using a seven-point Likert scale, ranging from 1 ("completely dissatisfied") to 7 ("delighted"). The scale will be explained to the patients and the total score will be calculated and recorded at the preoperative assessment (baseline) and at postoperative weeks 2, 4, 8, and 12.
Patient's activity level | 12 weeks postoperatively
  Postoperative Patient's activity level according to Barthel Activities of Daily Living scale (ADL).
  This scale comprises 10 basic daily activities (bowel, bladder, feeding, toilet, bathing, dressing, grooming, walking, stairs and transfer) with each item scored as 0 = need complete help, 1 = need some help or 2 = need no help
Total amount of morphine consumption | 48 hours postoperatively
  Rescue analgesia will be provided in the form of intravenous morphine 3 mg boluses if the patient indicates Visual Analogue Scale (VAS) ≥ 4.
Total amount of fentanyl consumption | Intraoperatively
  Rescue analgesia of fentanyl 1 μg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels.
Patient Global Impression of Change (PGIC) | 12 weeks postoperatively
  Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. PGIC is a 7-point scale depicting a patient's rating of overall improvement. 0 (very much worse" to 7 (very much improved).
Incidence of side effects of Pregabalin | 12 weeks postoperatively
  Side effects of Pregabalin such as headaches, feeling sleepy, tired or dizzy, diarrhoea, mood changes, feeling sick, swollen hands, arms, legs and feet, blurred vision, difficulties with getting an erection, and weight gain - because pregabalin can cause you feel hungry, and memory problems will be recorded.
Incidence of side effects of Pregabalin | 12 weeks postoperatively
  The side effects of Amantadine such as dry mouth, constipation, nausea, vomiting, decreased appetite, difficulty falling asleep or staying asleep, abnormal dreams, headache, confusion, drowsiness, tiredness, uncontrollable tightening of muscles, change from normal walking to falls, and a lace-like purple pattern on the skin.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author